CLINICAL TRIAL: NCT00819832
Title: Assessment of Circulating Tumor Cell Burden After Radiofrequency-Based Plasma Ablation (COBLATION®) in Conjunction With Vertebroplasty or Kyphoplasty for Augmenting Painful Vertebral Compression Fractures Secondary to Malignancy
Brief Title: Anderson Circulating Tumor Cell Burden (CTCB) Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated by sponsor.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: ArthroCare Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0593; NCT00756054 (obsolete NCT alias)
Record Dates: First submitted 2009-01-07; First posted 2009-01-09 (Estimated); Results first posted 2010-12-16 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Cancer; Spinal Disease; Vertebral Compression Fractures
Keywords: vertebral compression fractures; VCF; Spinal; Broken spinal bones; Kyphoplasty; vertebroplasty; Cavity SpineWand; Circulating Tumor Cell Burden; CTCB; Spine pain; Coblation; plasma radiofrequency ablation; Plasma-mediated ablation technology; precise molecular dissociation (ablation) process; medical cement
MeSH Terms: conditions — Neoplasms; Spinal Diseases | interventions — Kyphoplasty; Vertebroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Phase 1 Group 1 Vertebroplasty (Experimental): Vertebroplasty
  Interventions: Procedure: Vertebroplasty
- Phase 1 Group 2 Kyphoplasty (Experimental): Kyphoplasty
  Interventions: Procedure: Kyphoplasty
- Phase 2 Group 1 Vertebroplasty (Active Comparator): Vertebroplasty
  Interventions: Procedure: Vertebroplasty
- Phase 2 Group 2 Vertebroplasty + Cavity SpineWand (Active Comparator): Vertebroplasty with Cavity SpineWand
  Interventions: Procedure: Vertebroplasty; Device: Cavity SpineWand
- Phase 2 Group 3 Kyphoplasty (Active Comparator): Kyphoplasty
  Interventions: Procedure: Kyphoplasty
- Phase 2 Group 4 Kyphoplasty + Cavity SpineWand (Active Comparator): Kyphoplasty with Cavity SpineWand
  Interventions: Procedure: Kyphoplasty; Device: Cavity SpineWand

INTERVENTIONS:
Procedure: Kyphoplasty — A small fluid balloon will create a hole in the broken back bone where tumor is located. After balloon deflation and removal, hole is filled with medical cement.
  Arms: Phase 1 Group 2 Kyphoplasty; Phase 2 Group 3 Kyphoplasty; Phase 2 Group 4 Kyphoplasty + Cavity SpineWand
Procedure: Vertebroplasty — Medical cement will be injected into broken back bone.
  Arms: Phase 1 Group 1 Vertebroplasty; Phase 2 Group 1 Vertebroplasty; Phase 2 Group 2 Vertebroplasty + Cavity SpineWand
Device: Cavity SpineWand — Removes tissue (soft tissue, bone tissue, or both, but this will vary from person to person), including all or part of the cancerous tumors in the area of the broken back bone(s).
  Arms: Phase 2 Group 2 Vertebroplasty + Cavity SpineWand; Phase 2 Group 4 Kyphoplasty + Cavity SpineWand

SUMMARY:
Phase 1 - Optimization Phase:

Primary Objective: The primary objective of Phase 1 of this study is to determine the time point at which maximal Circulating Tumor Cell Burden (CTCB) occurs following standard vertebroplasty and Kyphoplasty procedures relative to baseline CTCB.

Phase 2 - Comparison Phase:

Primary Objective: The primary objective of Phase 2 of this study is to determine the change in CTCB from baseline to post-treatment as measured using the CellSearch™ Assay and to compare the average change between treatment groups with and without the use of the Cavity SpineWand.

Secondary Objectives:

* To determine the change in self-reported pain level from baseline to post-treatment as measured using the visual analogue scale (VAS) for spine pain and to compare the average change in pain level between treatment groups.
* To determine the change in pain status from baseline to post-treatment as measured using the Brief Pain Inventory (BPI) and to compare the average change in pain status between treatment groups.
* To determine the change from baseline to post-treatment in the M.D. Anderson Cancer Center Symptom Inventory (MDASI) and to compare the average change between treatment groups.
* To determine the change from baseline to post-treatment in time to walk a 50-foot distance and to compare the average change between treatment groups.

DETAILED DESCRIPTION:
Kyphoplasty and Vertebroplasty:

Kyphoplasty and vertebroplasty are types of surgery that are used to treat broken bones in the back, which may have been caused by cancer. Both procedures involve injecting a mixture of medical cement into the broken bone(s) in the back. The cement is designed to harden and become a permanent part of the bone, supporting the bone like an "internal cast" that brings it back to its original shape. The amount of cement will vary from person to person, but it could be, for example, anywhere from a fraction of a teaspoon to a full teaspoon.

The main difference between the 2 procedures is that kyphoplasty involves the use of a small medical type of balloon, and vertebroplasty does not use balloons. Vertebroplasty also uses a slightly smaller needle to inject the cement.

The Study Device:

The Cavity SpineWand is a rod-shaped surgical tool that is designed to use a type of energy called plasma in order to destroy tissue at lower temperatures than other surgical methods. This may help to lessen damage to other nearby tissue.

In this study, the Cavity SpineWand will be used to remove tissue (soft tissue, bone tissue, or both, but this will vary from person to person), including all or part of the cancerous tumors in the area of the broken bone(s). This is designed to make extra room for the cement to be injected, either during the vertebroplasty procedure or the kyphoplasty procedure.

Screening Tests:

Before you can receive treatment in this study, you will have "screening tests" to help the doctor decide if you are eligible to take part in this study. If you have had some of these tests done recently, they may not need to be repeated. This will be up to your study doctor. The following tests may be performed:

* Your medical history will be recorded.
* You will have a magnetic resonance imaging (MRI) scan and a computed tomography (CT) scan. These scans will show pictures of your broken back bone(s) and the tumor. Your doctor will use these pictures to plan your surgery.

Women who are able to have children must have a negative urine pregnancy test.

Doctors currently do not fully understand whether kyphoplasty or vertebroplasty is better for treating broken bones in the back. For this reason, and because this study involves randomly assigning participants to receive one or the other of these procedures, all participants must be eligible for both procedures in order to take part in this study.

Treatment Groups:

If you are found to be eligible to take part in the study, you will be assigned to a treatment group. In each phase of the study, there is an equal chance of being assigned to any of the treatment groups.

If you are one of the first 20 patients enrolled in the study, you will be enrolled in Phase 1. You will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. Phase 1 Group 1 will receive vertebroplasty, and Phase 1 Group 2 will receive kyphoplasty.

If you are one of the next 60 patients to be enrolled, you will be enrolled in Phase 2. You will be randomly assigned (as in the toss of dice) to 1 of 4 groups. Phase 2 Group 1 will receive vertebroplasty, and Phase 2 Group 2 will receive vertebroplasty with the Cavity SpineWand. Phase 2 Group 3 will receive kyphoplasty, and Phase 2 Group 4 will receive kyphoplasty with the Cavity SpineWand.

Study Tests/Procedures Before Surgery:

Within about 2-4 weeks before surgery, you will have tests and procedures performed. If you had some of these tests done recently, they may not need to be repeated. The following procedures may be performed:

* Your medical history will be recorded.
* You will have a physical exam, including measurement of vital signs (blood pressure, heart rate, temperature, and breathing rate).
* You will complete questionnaires that ask about the back pain and any drugs you are taking. In total, the questionnaires should take about 10-20 minutes to complete.
* You will be asked to walk 50 feet at your own pace while being timed to see how long it takes you. This is a routine test for comparing your walking function before and after surgery.

You will sign a separate consent form for surgery and the drugs used during surgery. These drugs include antibiotics to help lower the risk of infection, drugs to control pain, local anesthesia to make the area of your back where you are having surgery feel numb, and a sedative to make you feel relaxed and sleepy. The risks of these drugs will be explained to you in detail at that time.

Blood Test on the Day of Surgery:

On the day of surgery, blood (about 1 tablespoon) will be drawn. This blood will be compared with the blood that is drawn after surgery, to see when after surgery the most tumor cells are found in the blood.

Other Procedures Before Surgery:

As is standard for these types of surgery, special "bone" needles will be placed into the broken bone(s) in your back. X-rays will be used to guide the needles into a safe position. A biopsy of the tumor in your back bone will be collected to check the diagnosis of cancer. To collect a biopsy, a small amount of tumor tissue is withdrawn through the bone needle.

Surgical Procedures:

If you are in Phase 2 Group 2 or Phase 2 Group 4, the Cavity SpineWand will be used to remove a small amount of tissue immediately before the kyphoplasty or vertebroplasty procedure.

If you are in Phase 1 Group 2, Phase 2 Group 3, or Phase 2 Group 4, the kyphoplasty procedure will be done next. A small balloon will be placed into the area in your back where the tumor is located. Fluid will then be pumped through the tube in order to fill the balloon, which will create a hole in the back bone. After the balloon is deflated (closed) and removed, this hole will then be filled with cement. X-rays will be used to help place the cement safely.

If you are in Phase 1 Group 1, Phase 2 Group 1, or Phase 2 Group 2, the vertebroplasty procedure will be done next (instead of the kyphoplasty). Cement will be injected into the back bone. X-rays will be used to help place the cement safely.

No matter which treatment group you are in, if you have more than 1 broken back bone that needs treatment, the procedures described above will be repeated for a second broken bone, right after your first procedure. In other words, if you had vertebroplasty performed without the Cavity Spine Wand, that same procedure would be performed for the second bone. The procedure would only be repeated this 1 additional time, and not a third time.

No matter which treatment you receive, the entire procedure should take about 2-3 hours. If you need to have the procedure repeated on a second broken bone, this additional procedure should add about 45 minutes to the 2-3 hours that the first procedure alone would have taken.

Blood Testing for Phase 1 Participants:

Phase 1 participants will have blood (about 1 tablespoon each time) drawn at 8 different times points in order to measure the number of tumor cells. This blood will be drawn at 10, 30, and 60 minutes, and then at 2 hours, and between 6-8 hours, 10-18 hours, 20-28 hours, and 7 days after the surgery.

Blood Testing for Phase 2 Participants:

Phase 2 participants will have blood (about 1 tablespoon each time) drawn at 4 different time points after surgery. The first and second blood draw will occur before 36 hours has passed. The third blood draw will be about 36 hours after the surgery, and the fourth blood draw will be about 7 days after the surgery. This blood will be tested to measure the number of tumor cells.

Follow-Up Care:

You will be asked to return for follow-up visits at 7 days after your surgery and again at 4 weeks after your surgery. At these visits, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of vital signs.
* You will complete the questionnaires that ask about the back pain and any drugs you are taking.
* You will be asked to walk a 50-foot distance, and your walk will be timed.
* At the Day 7 visit only, blood (about 1 tablespoon) will be drawn to measure the number of tumor cells.
* At the Week 4 visit only, you will be asked to complete a questionnaire that asks you to rate how satisfied you feel with the surgery. It should take about 10 minutes to complete.

At 3 months after your surgery, the study staff will call you at home to ask about the back pain and any drugs you may be taking.

Length of Study Participation:

After the Month 3 follow-up phone call, your active participation in this study will be over. If it is determined after your surgery that the tumor in your back was not cancerous, you would still return for the follow-up visits as is standard, but you would not need to have the Day 7 blood test to measure the number of tumor cells.

This is an investigational study. The vertebroplasty and kyphoplasty procedures are commercially available and FDA approved for the way they are being used in this study. The Cavity SpineWand is also commercially available and FDA approved for the way it is being used in this study. The research-specific part of this study is the blood testing to measure any increases in the number of cancer cells in the blood.

Up to 100 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is >18 years old.
2. Patient is a candidate for standard vertebroplasty or Kyphoplasty with reasonable safety, as determined by the physician performing the procedure.
3. Patient is medically fit to undergo conscious sedation.
4. Patient is able to understand and give consent to participation in the study.
5. Patient presents with back pain >= 50 (on a 0-100 VAS scale).
6. Patient presents with a vertebral compression fracture believed to be due to malignancy.
7. Patient agrees to undergo, prior to the procedure, both magnetic resonance imaging (MRI, within 45 days of the planned procedure) and computed tomography (CT, within 14 days of the procedure). If MRI is contraindicated (due to pacemakers, intracranial ferromagnetic metal, etc), imaging with a nuclear medicine bone scan could be used as an alternative. CT remains mandated as a planning modality for all cases.
8. Patient has a life expectancy of at least 4 months.
9. Patient agrees to participate in the clinical study and to complete all required visits and evaluations.
10. Patient's vertebrae can safely be accessed with an 8 Gauge Cannula.
11. Suitable test for Circulating Tumor Cell Burden (CTCB) is available.

Exclusion Criteria:

1. Patient has unfavorable surgical anatomy to indicate that the patient could not be safely treated in any one of the four surgical groups if the patient was randomized to that group.
2. Patient has uncorrectable coagulopathy.
3. The metastatic lesions are determined to be blastic in nature and contain such sclerotic bone that the fracture site cannot adequately be accessed.
4. Vertebral compression fractures are present at multiple-levels and more than 2 levels must be treated during the same surgery (patients who have multi-level disease can still be enrolled provided no more than 2 levels be treated at one occasion).
5. Patient has significant risk of procedure-related complications due to potential interactions with devices or materials used in the procedures, i.e., Pacemaker implant or Allergy (e.g., to cement, cannula metal, contrast medium, etc.)
6. Patient is unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawid Schellingerhout, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: December 30, 2008 to March 29, 2010. All recruitment done at UT MD Anderson Cancer Center.
Pre-assignment Details: Study terminated by sponsor. No patient data analysis performed due to the limited amount of data gathered from the study's three participants.
Groups:
- Phase 2 Group 2 Vertebroplasty +Cavity SpineWand: Vertebroplasty with Cavity SpineWand
Period: Overall Study
Arm/Group | Phase 1 Group 1 Vertebroplasty | Phase 1 Group 2 Kyphoplasty | Phase 2 Group 1 Vertebroplasty | Phase 2 Group 2 Vertebroplasty +Cavity SpineWand | Phase 2 Group 3 Kyphoplasty | Phase 2 Group 4 Kyphoplasty + Cavity SpineWand
Started | 3 (No patient data analysis.) | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Termination of Study | 3 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Group 1 Vertebroplasty | Phase 1 Group 2 Kyphoplasty | Phase 2 Group 1 Vertebroplasty | Phase 2 Group 2 Vertebroplasty +Cavity SpineWand | Phase 2 Group 3 Kyphoplasty | Phase 2 Group 4 Kyphoplasty + Cavity SpineWand | Total
Number analyzed (Participants) | 3 | 0 | 0 | 0 | 0 | 0 | 3
Age, Continuous [Median (Full Range); unit: years] | 63 [49 to 75] |  |  |  |  |  | 63 [49 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 |  |  |  |  |  | 3
  Male | 0 |  |  |  |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 |  |  |  |  |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Time to Maximal Circulating Tumor Cell Burden (CTCB)
Description: Increase in number of cancer cells in patient's blood after standard kyphoplasty or vertebroplasty treatment of broken back bones that may have been caused by cancer measured by CTCB evaluation from peripheral blood (10cc) collected at 8 varying time points for a total of 100 cc collected over the 7 day period of time (10, 30, and 60 minutes, and then at 2 hours, and between 6-8 hours, 10-18 hours, 20-28 hours, and 7 days after the surgery).
Time Frame: Pre-procedure baseline blood draws through post surgery 24 hours followed at 7 days (+/- 2 days)
Population: Study terminated by sponsor; No data analysis done on limited amount of data gathered.
Arm/Group | Phase 1 Group 1 Vertebroplasty | Phase 1 Group 2 Kyphoplasty | Phase 2 Group 1 Vertebroplasty | Phase 2 Group 2 Vertebroplasty +Cavity SpineWand | Phase 2 Group 3 Kyphoplasty | Phase 2 Group 4 Kyphoplasty + Cavity SpineWand
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Phase 2: Change in CTCB From Baseline to Post-treatment
Time Frame: CTCB evaluation performed from baseline through surgery +24 hours to post 7 days (+/- 2 days)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 15 months
Description: No patients were enrolled in other groups or Phase II.
Arm/Group | Phase 1 Group 1 Vertebroplasty | Phase 1 Group 2 Kyphoplasty | Phase 2 Group 1 Vertebroplasty | Phase 2 Group 2 Vertebroplasty +Cavity SpineWand | Phase 2 Group 3 Kyphoplasty | Phase 2 Group 4 Kyphoplasty + Cavity SpineWand
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No